CLINICAL TRIAL: NCT02633566
Title: Randomized Clinical Trial of the Effect of Functional Orthoses on the Joint Position of the Hindfoot in Children With Flat Feet After a Year of Follow-up
Brief Title: Clinical Trial of the Effect of Functional Orthoses in Children With Flat Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresno, Raquel Lopez, M.D. (Individual)
Responsible Party: Principal Investigator, Raquel Lopez Fresno, PhD Student (Podiatrist), Fresno, Raquel Lopez, M.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Flexible Flatfoot
Keywords: Flatfoot; orthoses; children
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional plantar orthoses (Active Comparator): Functional plantar orthoses in polypropylene with Medial Heel Skive technique
  Interventions: Device: Plantar orthoses
- Placebo plantar orthoses (Placebo Comparator): Plantar orthoses made in Ethil Vinyl Acetate (22º Shore) without correction of the pronation
  Interventions: Device: Plantar orthoses

INTERVENTIONS:
Device: Plantar orthoses

SUMMARY:
The purpose of this study is to investigate the efficay of functional plantar orthoses on flatfoot in children.

DETAILED DESCRIPTION:
There's a considerable controversy regarding the effectiveness of plantar orthoses in the treatment of flexible flat foot, despite being the most widely used treatment. Several studies tried to investigate the correction of the deformity using plantar orthoses, but there are few studies with a control group of people, not enough to compare the effectiveness of the treatment.

A randomized, double-blind, parallel design clinical trial was conducted with two study groups. The sample consisted of 61 children, aged 3 and 4 years old, who were randomly assigned to each study group. One group (intervention group) received treatment with functional plantar orthotics, and the other group (control group) received treatment with placebo-type plantar orthotics, to use as a reference or comparison. Both groups were followed for a one-year period. Before delivering the treatment, all subjects underwent dorsoplantar radiography, repeated at the end of the treatment (after one year). Differences in the talus-calcaneus, tibionavicular and talus-first metatarsal angles were compared, pre and post-treatment of both study groups. Test analysis of covariance (ANCOVA) was performed as a statistical test.

ELIGIBILITY:
Inclusion Criteria:

* Flexible flatfoot

Exclusion Criteria:

* Congenital Vertical talus
* Tarsal coalition
* Neuromuscular disease
* Ligamentous laxity
* Previous history of surgery on lower limb
* Previous orthotic treatment

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
X-ray measurements of the angles: talus-calcaneus, talus-navicular and talus-first metatarsal angle. | One year
  Before delivering the treatment, all subjects underwent dorsoplantar radiography, repeated at the end of the treatment (after one year). Differences in the talus-calcaneus, tibionavicular and talus-first metatarsal angles were compared, pre and post-treatment of both study groups. Test analysis of covariance (ANCOVA) was performed as a sataistical test.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pascual Huerta, PhD, Study Director

REFERENCES:
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub4. PMID 35080267
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 14;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub3. PMID 35029841